CLINICAL TRIAL: NCT01808534
Title: Multicenter Single Arm Phase II Study of Single Agent Palifosfamide in Recurrent and Incurable Germ Cell Tumors
Brief Title: Palifosfamide in Treating Patients With Recurrent Germ Cell Tumors
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Due to Low Accrual
Sponsor: Indiana University School of Medicine (Other)
Collaborators: Alaunos Therapeutics (Industry)
Responsible Party: Sponsor
Organization: Indiana University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IUCRO-0403; NCI-2013-00510 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 1301010501 (Other: Indiana University Institutional Review Board)
Record Dates: First submitted 2013-03-06; First posted 2013-03-11 (Estimated); Results first posted 2015-07-02 (Estimated); Last update posted 2015-07-02 (Estimated); Status verified 2015-06

CONDITIONS: Adult Central Nervous System Germ Cell Tumor; Adult Teratoma; Malignant Extragonadal Germ Cell Tumor; Malignant Extragonadal Non-Seminomatous Germ Cell Tumor; Extragonadal Seminoma; Recurrent Malignant Testicular Germ Cell Tumor; Recurrent Ovarian Germ Cell Tumor; Stage IV Extragonadal Non-Seminomatous Germ Cell Tumor; Stage IV Extragonadal Seminoma; Stage IV Ovarian Germ Cell Tumor
MeSH Terms: conditions — Teratoma; Testicular Neoplasms | interventions — isophosphamide mustard; Ifosfamide; palifosfamide lysine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (palifosfamide) (Experimental): Patients receive palifosfamide IV over 30 minutes on days 1-3. Treatment repeats every 21 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: palifosfamide

INTERVENTIONS:
Drug: palifosfamide — Given IV
  Other Names: IPM-lysine; isophosphoramide mustard-lysine; ZIO-201

SUMMARY:
This phase II trial studies how well palifosfamide works in treating patients with recurrent germ cell tumors. Drugs used in chemotherapy, such as palifosfamide, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the response rate (complete response [CR]+partial response [PR]) of single agent palifosfamide in patients with refractory germ cell tumors.

SECONDARY OBJECTIVES:

I. To determine the duration of remission. II. To determine progression free and overall survival. III. To assess toxicity and tolerability of palifosfamide in patients with germ cell tumors.

OUTLINE:

Patients receive palifosfamide intravenously (IV) over 30 minutes on days 1-3. Treatment repeats every 21 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months for 3 years, every 6 months for 2 years, and then annually thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histological or serological proof of metastatic germ cell neoplasm (gonadal or extragonadal primary) with disease not amenable to cure with either surgery or chemotherapy; patients with seminoma and nonseminoma are eligible, as are women with ovarian germ cell tumors
* Patients must have evidence of recurrent or metastatic carcinoma by one or more of the criteria specified in the protocol
* Patients must have received initial cisplatin based combination therapy (such as bleomycin, etoposide and cisplatin [BEP], etoposide and cisplatin [EP], VP-16 plus ifosfamide plus cisplatin [VIP] or similar regimens) AND demonstrated progression following the administration of at least one 'salvage' regimen for advanced germ cell neoplasm (such as high dose chemotherapy, paclitaxel/ifosfamide/cisplatin [TIP] or vinblastine, ifosfamide and cisplatin [VeIP])
* Patients must have documented "failure" of prior therapy as defined in the protocol
* Patients are eligible after first line platinum based chemotherapy if their disease has relapsed and they have primary mediastinal non seminomatous germ cell tumor (PMNSGCT) or late relapse (> 2 years) not amenable to surgical resection
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Laboratory test results must be within ranges established in the protocol
* Potential subject must have the ability to understand (as judged by the treating physician) and willingness to provide written informed consent and Health Insurance Portability and Accountability Act (HIPAA) authorization for release of personal health information;
* Females of childbearing potential must not be pregnant or breast-feeding; male and female patients of reproductive potential must agree to use a highly reliable method of birth control from the screening visit through 28 days after the last dose of study drug

Exclusion Criteria:

* No active clinically serious infections as judged by the treating investigator (> CTCAE grade 2) including known human immunodeficiency virus (HIV) infection or chronic active hepatitis B or active hepatitis C
* No presence of, or history of any illness or injury to the urinary tract which may make the patient more susceptible to acute renal insufficiency in the case of potential renal adverse events
* Patients must not have any cardiac disorders as defined in the protocol
* No history of psychiatric illness/social situations that would limit compliance with study requirements
* Patients must be at least 4 weeks post major surgery or significant traumatic injury at time of study registration
* Patients must be at least 7 days post any minor surgical procedure, excluding placement of a vascular access device at the time of study registration
* Patients must not have a known sensitivity to any component of palifosfamide or its known excipients
* Patients with active central nervous system (CNS) metastases are excluded
* Patients must not have previously been exposed to palifosfamide
* Patients must have at least 3 weeks after previous radiotherapy or chemotherapy and have recovered from all major toxicities (except alopecia or grade 1 or 2 neuropathy) at the time of registration

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2013-02; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence H Einhorn, MD, Principal Investigator — Indiana University School of Medicine
Locations (3):
- United States (3):
  - Indiana University Cancer Center, Indianapolis, Indiana
  - Abramson Cancer Center of The University of Pennsylvania, Philadelphia, Pennsylvania
  - Virginia Mason Medical Center, Seattle, Washington

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This protocol was based on a two stage design, getting 12 patients at the first stage and 8 more if at least one CR or PR was observed in the first 12. Due to low accrual, the study was stopped at 5 patients for this study.
Period: Overall Study
Arm/Group | Treatment (Palifosfamide)
Started | 5
Completed | 1
Not Completed | 4
Not completed — Disease progression | 3
Not completed — Physician Decision | 1

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Palifosfamide)
Number analyzed (Participants) | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 5
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.6 (13.83)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 4
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 4
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate (Defined as Partial Response or Complete Response)
Description: The percent of patients who were shown as having a partial remission or better based on definitions of response in RECIST 1.1. At least a 30% decrease in the sum of the diameters of target lesions, in reference to baseline sum diameters, needs to be confirmed to be considered as partial response or better. Note: There were no patients with a partial or complete response.
Time Frame: Up to 2 years
Population: All patients who enrolled and received treatment with at least one post baseline assessment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment (Palifosfamide)
Number analyzed (Participants) | 5
percentage of participants | 0 [0 to 0]

2. Secondary Outcome: Duration of Remission in Patients Who Achieve a Partial or Complete Response
Description: The duration of remission is from the time of confirmed partial or complete response until progression or death. Patients continuing in remission at the end of the study will be treated as censored. Summarized by Kaplan-Meier methods including 90% confidence intervals for the median using method of Brookmeyer and Crowley. Note: There were no patients who achieved partial or complete response.
Time Frame: Up to 2 years
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | Treatment (Palifosfamide)
Number analyzed (Participants) | 5
months | 0 [0 to 0]

3. Secondary Outcome: Progression Free Survival (PFS)
Description: Summarized by Kaplan-Meier methods including 90% confidence intervals for the median using method of Brookmeyer and Crowley. Time until progression, death or last evaluation will be calculated. If a patient did not progress or die, they will be censored at their last evaluation in the analysis.
Time Frame: Up to 2 years
Population: All patients who enrolled and received treatment.
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | Treatment (Palifosfamide)
Number analyzed (Participants) | 5
months | 0.69 [0.07 to 6.18]

4. Secondary Outcome: Overall Survival
Description: Summarized by Kaplan-Meier methods including 90% confidence intervals for the median using method of Brookmeyer and Crowley. Time until death or last evaluation will be calculated. If a patient did not die, they will be censored in the analysis at their last known alive date.
Time Frame: Up to 2 years
Population: All patients who enrolled and received treatment.
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | Treatment (Palifosfamide)
Number analyzed (Participants) | 5
months | 0.95 [0.56 to 15.63]

5. Secondary Outcome: Treatment Related Adverse Events Grade 3 or Higher
Description: Number of unique patients who had a treatment related (possible, probable or definite) adverse event that was graded 3 or greater according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) v4.03.
Time Frame: Up to 2 years
Population: All patients who enrolled and received treatment.
Measure: Number; unit: participants
Arm/Group | Treatment (Palifosfamide)
Number analyzed (Participants) | 5
participants | 1

ADVERSE EVENTS:
Time Frame: Up to 2 years
Arm/Group | Treatment (Palifosfamide)
Serious Adverse Events (participants affected / at risk) | 2/5
Other Adverse Events (participants affected / at risk) | 4/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Palifosfamide) (N=5)
Small intestinal obstruction (Gastrointestinal disorders) | 1
Hypoglycemia (Metabolism and nutrition disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Palifosfamide) (N=5)
Abdominal pain (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 3
Diarrhea (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 2
Edema limbs (General disorders) | 1
Fatigue (General disorders) | 4
Non-cardiac chest pain (General disorders) | 1
Pain (General disorders) | 1
Anorexia (Metabolism and nutrition disorders) | 2
Back pain (Musculoskeletal and connective tissue disorders) | 2
Peripheral sensory neuropathy (Nervous system disorders) | 1
Insomnia (Psychiatric disorders) | 1
Acute kidney injury (Renal and urinary disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1
Thromboembolic event (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes